CLINICAL TRIAL: NCT06371261
Title: Pathogenicity of Species of the Achromobacter Genus in Patients With Cystic Fibrosis: a Prospective Multicentre Exploratory Study of a Cohort in Réunion Island.
Brief Title: Pathogenicity of Species of the Achromobacter Genus in Patients From Reunion Island With Cystic Fibrosis
Acronym: ACHROMO-MUCO
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/CHU/07
Record Dates: First submitted 2024-04-02; First posted 2024-04-17 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Cystic Fibrosis
Keywords: Achromobacter species; MALDI-TOF mass spectrometry; Réunion Island
MeSH Terms: conditions — Cystic Fibrosis | interventions — Biological Oxygen Demand Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Biological analyses — A cytobacteriological examination of the sputum will be carried out and sent to the microbiology laboratory at the University Hospital of La Réunion.
  The micro-organisms will be quantified.
  The micro-organisms, and more specifically bacteria of the Achromobacter genus, will be identified by MALDI-TOF mass spectrometry using the published database (Garrigos et al.2021).

SUMMARY:
The pathogenicity of Achromobacter bacteria is not yet well established, but studies show a decline in respiratory function and an increase in mortality associated with chronic colonisation, making it possible to classify the Achromobacter genus as an emerging pathogen in cystic fibrosis. It is possible that certain species or clones are more virulent or resistant, requiring the adaptation of measures to prevent cross-transmission in the centres concerned.

However, until now, the identification of Achromobacter species has involved the use of molecular biology techniques that are not routinely applicable in diagnostic laboratories, limiting studies and the collection of epidemiological data. Recently, a database using MALDI-TOF mass spectrometry has been built for rapid and accurate species identification.

In view of the local epidemiology and the current lack of data, it would be necessary and interesting to use this tool to study a cohort of cystic fibrosis patients in Réunion island (North and South sites) to see whether one species has a greater clinical impact than another (pathogenicity), and/or is more responsible for chronic colonisation.

DETAILED DESCRIPTION:
The research hypotheses are: What is the pathogenicity of Achromobacter species in cystic fibrosis patients? Is the pathogenicity of one species of the genus Achromobacter greater than that of other species in cystic fibrosis patients, depending on the colonization status of this bacterial species? Colonization with a species of the genus Achromobacter is associated with an increased frequency of pulmonary exacerbations in cystic fibrosis patients.

Investigator will therefore assess the frequency of pulmonary exacerbations as a function of the Achromobacter species colonizing/infecting cystic fibrosis patients.

As this is an exploratory study carried out mainly on bacterial strains from patients, it presents no risk to patients.

the results of the study will enable clinicians to improve their knowledge of the different species of bacteria in the Achromobacter genus, in terms of pathogenicity, ability to colonize the respiratory tract, resistance and virulence.

As far as patients are concerned, the knowledge gained from this study will help improve the overall management of their disease. It will also provide food for thought on the establishment of guidelines and recommendations for dealing with Achromobacter spp. colonization and therapeutic strategy.

ELIGIBILITY:
Inclusion Criteria:

* Minor or major cystic fibrosis patients
* Patients with at least one sputum cytobacteriological test positive for Achromobacter spp. during the inclusion period.
* Patients living in La Réunion island.
* Patients for whom a non-opposition was obtained orally (if applicable from both one of the child's legal guardians and the child him/herself)

Exclusion Criteria:

* Patients without cystic fibrosis.
* Patients with cystic fibrosis but no Achromobacter-positive ECBC during the study inclusion period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohort of cystic fibrosis patients from Reunion island with Achromobacter spp colonisation
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Frequency of pulmonary exacerbations according to the species of the Achromobacter genus colonising/infecting cystic fibrosis patients. | 2 years
  The occurrence of pulmonary exacerbations as a function of the species of the genus Achromobacter spp. Colonising/infecting patients.

SECONDARY OUTCOMES:
Frequency of pulmonary exacerbations as a function of Achromobacter spp. colonisation status. | 2 years
  The occurrence of pulmonary exacerbations according to the colonisation statuses defined according to the French National Diagnostic and Care Protocol (PNDS)-Mucoviscidose of the French National Authority for Health (HAS) July 2017.
Emergence or existing presence of clones within the species of the genus Achromobacter circulating among cystic fibrosis patients in Réunion, using genomic analyses. | 2 years
  Clonality between strains: whole genome sequencing with genotyping between strains
Presence of virulence factors in these strains using genomic analyses | 2 years
  Study of the virulome: whole genome sequencing in search of virulence genes
Search for genes responsible for antibiotic resistance by genomic analysis of these strains | 2 years
  Study of the resistome: whole genome sequencing in search of resistance genes, antibiotic sensitivity tests
To describe the epidemiology of Achromobacter spp. in cystic fibrosis patients in Réunion | 2 years
  Prevalence of chronic colonisation with Achromobacter spp. and prevalence of colonisation according to Achromobacter species

CONTACTS AND LOCATIONS:
Overall Officials: Thomas GARRIGOS, Pharm D, PhD, Study Director — CHU La Réunion
Locations (2):
- Reunion (2):
  - CHU la Réunion North, Saint-Denis
  - CHU la Réunion South, Saint-Pierre

IPD SHARING:
Plan to Share IPD: No